CLINICAL TRIAL: NCT02881060
Title: The Late Effects of Ethanol Intake on the Glucose Response to Subcutaneous Glucagon in Type 1 Diabetes
Acronym: ALCO1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Danish Diabetes Academy (Other); University of Copenhagen (Other)
Responsible Party: Principal Investigator, Ajenthen Ranjan, MD, PhD student, Hvidovre University Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: H-16027080
Record Dates: First submitted 2016-08-11; First posted 2016-08-26 (Estimated); Last update posted 2017-07-24 (Actual); Status verified 2017-07

CONDITIONS: Hypoglycemia; Diabetes Mellitus, Type 1
Keywords: Glucagon; Ethanol
MeSH Terms: conditions — Hypoglycemia; Diabetes Mellitus, Type 1 | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ethanol (Active Comparator): Drinking a cocktail of ethanol (0.8 g ethanol per kg body weight), diet lemonade and water of 1:1:1 (volume distribution).
  Interventions: Dietary Supplement: Alcohol
- Non-ethanol (Placebo Comparator): Drinking a cocktail of diet lemonade and water of 1:2 (volume distribution).
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Alcohol
  Other Names: Cocktail
  Arms: Ethanol
Dietary Supplement: Placebo
  Other Names: Mocktail
  Arms: Non-ethanol

SUMMARY:
Objective: Because many people with type 1 diabetes drink ethanol and because glucagon is used to treat mild hypoglycaemia, it is essential to determine whether ethanol will impair the effectiveness of glucagon to increase glucose, which may impair the effectiveness of the dual hormone treatment in preventing hypoglycaemia.

The purpose of this study is to determine, whether ethanol influences the glucose response to subcutaneous glucagon during mild hypoglycaemia.

The investigators hypothesize that prior evening ethanol consumption does not reduce the effect of a glucagon bolus to raise plasma glucose compared with no prior ethanol consumption.

The study aims:

1. To determine the late effects of ethanol on the efficacy of subcutaneous glucagon to restore plasma glucose after an episode of mild hypoglycemia.
2. To determine the late effects of ethanol on the counter-regulatory hormones and hypoglycaemia awareness during mild hypoglycaemia

A double-blinded placebo-controlled study will be conducted. Participants will serve as their own controls. Eligible participants will after an informed consent complete two study visits, one with and one without ethanol consumption, in a random order. On each study visit, participants are induced a insulin induced hypoglycemia, seven-eight hours after a meal with or without ethanol. Once plasma glucose is below 3.9 mmol/l, a subcutaneous injection of 100 mcg glucagon is administered. Two hours later a second bolus is administered.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 70 years
* T1D ≥ 3 year
* BMI 20-28 kg/m2
* CSII ≥ 1 year
* Caucasian origin
* Hypoglycaemia awareness (assessed by Gold, Clarke and Pedersen-Bjergaard methods)
* Use of carbohydrate counting and the insulin pump bolus calculator for all meals
* Ethanol exposure once within 1 year consisting of at least 4 drinks (1 drink contains 12 gram ethanol) within four hours

Exclusion Criteria:

* Allergy or intolerance to lactose or Glucagen®(Novo Nordisk, Bagsværd, DK)
* Allergy for ethanol or any food ingredients that will be used in the study.
* Impaired renal function (eGFR < 60 ml/min/1.73m2)
* Liver disease with ALAT > 2.5 times the upper limit of the reference interval
* Gastropareses (beat-beat variation < 10 beats per min and/or orthostatic systolic blood pressure > 20 mmHg)
* Insomnia, sleep apnoea or any troubles with sleeping that according to the investigator's assessment makes the individual unsuitable for study participation.
* Aldehyde dehydrogenase deficiency as determined by a screening questionnaire
* Unable to refrain from the consumption of ethanol at least 24 hours prior to study start
* History of drinking problems or alcoholism, regardless of whether active or in remission.
* Use of benzodiazepines or barbiturates or opiates or other central nervous system depressant drugs that could act synergistically with ethanol to lower the level of consciousness
* History of drug abuse
* Current participation in another diabetes-related clinical trial that, in the judgment of the principle investigator, will compromise the results of the study or the safety of the subject.
* Use of anti-diabetic medicine (other than insulin), corticosteroids or other drugs affecting glucose metabolism during the study period or within 30 days prior to study start
* Use of medications that are known to cause QT interval prolongation
* Presence of pheochromocytoma
* Other concomitant medical or psychological condition that according to the investigator's assessment makes the individual unsuitable for study participation
* Females who are pregnant, breast-feeding or intend to become pregnant or are not using adequate contraceptive methods.
* Females who have different basal insulin pattern depending on their menstrual cycle.
* Inability to understand the individual information and to give informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-08; Primary Completion 2017-01-26 (Actual); Study Completion 2017-01-26 (Actual)

PRIMARY OUTCOMES:
Increase in plasma glucose | 0-120 min after the first glucagon injection
  The primary endpoint is difference in increase in plasma glucose value after the first injection of 100 µg s.c. glucagon on study nights with ethanol vs. study nights without ethanol consumption.

SECONDARY OUTCOMES:
Peak plasma glucose | 0-240 min after the first glucagon injection
  Maximal plasma glucose after the first and second glucagon injection
Increase in plasma glucose | 0-120 min after the second glucagon injection
  Increase in plasma glucose caused by the second glucagon injection.
Total AUC(0-120) | 0-240 min after the first glucagon injection
  Total area under the glucose curve from 0-120 minutes after each glucagon injection
PI-AUC(0-120) | 0-240 min after the first glucagon injection
  positive incremental area under the glucose curve from 0-120 minutes after each glucagon injection
Tmax | 0-240 min after the first glucagon injection
  Time-to-peak glucose value after each glucagon injection glucagon injection
Time above 4.0mM | 0-240 min after the first glucagon injection
  Duration of glucose above 4.0 mmol/l after first and second glucagon injection
Time above baseline | 0-240 min after the first glucagon injection
  Duration of glucose above baseline after first and second glucagon injection
Rescue rates | 0-240 min after the first glucagon injection
  Numbers of first and second glucagon injections that raises PG > 4.9 mmol/l
Hyperglycemia rates | 0-240 min after the first glucagon injection
  Number of first and second glucagon injections that raises PG > 7.1 mmol/l
Changes in plasma ketone bodies, measured as area under the curve | 0-240 min after the first glucagon injection
Changes in plasma ketone bodies, measured as incremental peak | 0-240 min after the first glucagon injection
Changes in plasma glucagon, measured as area under the curve | 0-240 min after the first glucagon injection
Changes in plasma glucagon, measured as incremental peak | 0-240 min after the first glucagon injection
Changes in insulin, measured as area under the curve | 0-240 min after the first glucagon injection
Changes in insulin, measured as incremental peak | 0-240 min after the first glucagon injection
Changes in growth hormones, measured as area under the curve | 0-240 min after the first glucagon injection
Changes in growth hormones, measured as incremental peak | 0-240 min after the first glucagon injection
Changes in serum corticole, measured as area under the curve | 0-240 min after the first glucagon injection
Changes in serum corticole, measured as incremental peak | 0-240 min after the first glucagon injection
Changes in plasma ethanol, measured as area under the curve | 0-240 min after the first glucagon injection
Changes in plasma ethanol, measured as incremental peak | 0-240 min after the first glucagon injection
Changes in free fatty acids, measured as area under the curve | 0-240 min after the first glucagon injection
Changes in free fatty acids, measured as incremental peak | 0-240 min after the first glucagon injection
Changes in triglycerides, measured as area under the curve | 0-240 min after the first glucagon injection
Changes in triglycerides, measured as incremental peak | 0-240 min after the first glucagon injection
Average in blood pressure | 0-240 min after the first glucagon injection
Average heart rate | 0-240 min after the first glucagon injection
Intensity of hypoglycemia | 0-240 min after the first glucagon injection
  Average changes in Edinburgh Hypoglycaemia Scale over time during insulin and glucagon phase
Cognitive impairment | 0-240 min after the first glucagon injection
  Average scores in cognitive test 30 min before each glucagon injection.
Side effects | 0-240 min after the first glucagon injection
  Average visual analogue scale score from 0-180 min for nausea and headache after glucagon injection
Incidence of vomiting | 0-240 min after the first glucagon injection
  Incidence of vomiting after 0-4 hours after each glucagon injection.
Meal induced glucose excursion | 0-3 hours after meal
  Total and incremental area under the glucose curve from 0-120 and 0-240 min after eating the mixed meal
Meal induced hormonal changes | 0-3 hours after meal
  Total and incremental area under the glucose curve from 0-120 and 0-240 min after eating the mixed meal
Nocturnal changes in plasma glucose | 0-6 hours after start of sleep
  Area under the curve during sleep
Nocturnal changes in corticol | 0-6 hours after start of sleep
  Area under the curve during sleep
Nocturnal changes in growth hormone | 0-6 hours after start of sleep
  Area under the curve during sleep
Nocturnal changes in ketones | 0-6 hours after start of sleep
  Area under the curve during sleep
Nocturnal changes in ethanol | 0-6 hours after start of sleep
  Area under the curve during sleep
Nocturnal changes in glucagon | 0-6 hours after start of sleep
  Area under the curve during sleep
Difference between the first second glucagon injection and between both study visits in peak change plasma glucose | 0-240 min after the first glucagon injection
Difference between glucagon injections on both study visits in positive incremental area under the glucose curve from 0-120 minutes | 0-240 min after the first glucagon injection
Difference between glucagon injections on both study visits in total area under the glucose curve from 0-120 minutes | 0-240 min after the first glucagon injection
Difference between glucagon injections on both study visits in time-to-peak glucose value | 0-240 min after the first glucagon injection
Difference between glucagon injections on both study visits in duration of glucose above 4.0 mmol/l after first and second glucagon injection | 0-240 min after the first glucagon injection
Difference between glucagon injections on both study visits in duration of glucose above baseline after first and second glucagon injection | 0-240 min after the first glucagon injection
Difference in glucose sensor data on study night with alcohol vs. study night without alcohol - Mean absolute relative difference (MARD) values of glucose sensors compared with YSI from 7 PM- 8 AM. | 0-10 hours after meal
  Intentions to treat analysis
Difference in glucose sensor data on study night with alcohol vs. study night without alcohol - Precision absolute relative difference (PARD) 120 min before and 120 after each glucagon injection. | 0-10 hours after meal
  Intentions to treat analysis
Difference in glucose sensor data on study night with alcohol vs. study night without alcohol - MARD values between glucose sensors 0-120 minutes after each glucagon injection. | 0-10 hours after meal
  Intentions to treat analysis
Difference in glucose sensor data within 2 days after study night with alcohol vs. study night without alcohol - Time in range (glucose sensor value =4.0-10.0mmol/l) | 0-2 days after the first glucagon injection
  Intentions to treat analysis
Difference in glucose sensor data within 2 days after study night with alcohol vs. study night without alcohol - Time in hypoglycaemia (glucose sensor value < 4.0 mmol/l) | 0-2 days after the first glucagon injection
  Intentions to treat analysis
Difference in glucose sensor data within 2 days after study night with alcohol vs. study night without alcohol - Time in hyperglycaemia (glucose sensor value >10.0mmol/l) | 0-2 days after the first glucagon injection
  Intentions to treat analysis
Difference in glucose sensor data within 2 days after study night with alcohol vs. study night without alcohol - Number of hypoglycaemia episodes (glucose sensor value < 4.0 mmol/l) | 0-2 days after the first glucagon injection
  Intentions to treat analysis
Difference in glucose sensor data between the study period with and without alcohol - Clarke- Error Grid analysis for both sensors compared with YSI during study visit | -2 to 4 days after study visits
  Intentions to treat analysis
Difference in glucose sensor data between the study period with and without alcohol - PARD values from day 1-7 | -2 to 4 days after study visits
  Intentions to treat analysis
Difference in glucose sensor data between the study period with and without alcohol - PARD values <4.0 mmol/L from day 1-7 | -2 to 4 days after study visits
  Intentions to treat analysis
Difference in glucose sensor data between the study period with and without alcohol - PARD values 4.0-10.0 mmol/L from day 1-7 | -2 to 4 days after study visits
  Intentions to treat analysis
Difference in glucose sensor data between the study period with and without alcohol PARD values >10.0 mmol/L from day 1-7 | -2 to 4 days after study visits
  Intentions to treat analysis
Difference in glucose sensor data between the study period with and without alcohol - Number of hypoglycaemia episodes (glucose sensor value < 4.0 mmol/l) | -2 to 4 days after study visits
  Intentions to treat analysis

CONTACTS AND LOCATIONS:
Overall Officials: Ajenthen Ranjan, MD, Principal Investigator — Hvidovre University Hospital
Locations (1):
- Hvidovre University Hospital, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: Undecided